CLINICAL TRIAL: NCT06838728
Title: The Effect of the Application of Head Mounted Magnifying Glasses on Postoperative PTH Changes in Thyroid Surgery: Stage II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Collaborators: Second Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Guojun Wu, chief physician, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SWYX2024-280
Record Dates: First submitted 2025-02-15; First posted 2025-02-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Surgery
Keywords: thyroid cancer; thyroid surgery; Head Mounted Magnifying Glasses
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: This study was divided into an experimental group and a control group based on whether a head mounted magnifying glass was used, with the main calculation indicator being changes in PTH levels before and after surgery.
Who Masked: Participant, Outcomes Assessor
Masking Description: no other parties
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): When the experimental group undergoes surgery, the surgeon uses a head mounted magnifying glass to assist in the surgical operation.
  Interventions: Device: Head Mounted Magnifying Glasses
- control group (No Intervention): When the experimental group undergoes surgery, the surgeon don't use a head mounted magnifying glass to assist in the surgical operation.

INTERVENTIONS:
Device: Head Mounted Magnifying Glasses — This study was divided into an experimental group and a control group based on whether a head mounted magnifying glass was used.
  Arms: experimental group

SUMMARY:
This study is a prospective research. This study aims to investigate and follow up patients who undergo open thyroidectomy in the Department of Breast and Thyroid Surgery at Shandong Provincial Hospital from January 2020 to December 2025. This study was divided into an experimental group and a control group based on whether a head mounted magnifying glass was used, with the main calculation indicator being changes in PTH levels before and after surgery. This study investigated whether the application of head mounted magnifying glasses had an impact on preoperative and postoperative changes in PTH levels through inter group and self pre - and post control, in order to verify the practical effectiveness of head mounted magnifying glasses in thyroid surgery and provide reasonable suggestions for the selection of subsequent surgical treatment methods.

DETAILED DESCRIPTION:
In thyroid surgery, changes in postoperative parathyroid hormone (PTH) levels have a significant impact on the patients recovery and long-term health status. Parathyroid hormone is responsible for regulating blood calcium levels, and its dysfunction can cause serious electrolyte imbalance and metabolic problems. In the process of thyroid surgery, especially in total thyroidectomy, protecting the function of the parathyroid gland is an important operation. The diameter of the parathyroid gland is small and similar to the morphology of lymph nodes, making it susceptible to damage during surgery. Although traditional magnification tools such as surgical microscopes have certain effects, their operation is complex and their adaptability to surgical scenes is limited.

In recent years, as an emerging magnifying tool, head mounted magnifying glasses have been increasingly used in thyroid surgery due to their portability, ease of operation, and providing a larger field of view. Wearing a head mounted magnifying glass can not only improve the clarity of vision during surgery, increase the recognition rate of parathyroid glands and nerves, but also reduce the risk of parathyroid injury by improving surgical accuracy, thereby more effectively maintaining the stability of postoperative PTH levels. In addition, the use of head mounted magnifying glasses can reduce surgical time, intraoperative uncertainty, and the risk of postoperative complications.

This study systematically evaluates the changes in PTH levels before and after surgery to verify the practical effectiveness of head mounted magnifying glasses in thyroid surgery, and further explores the effectiveness of parathyroid gland protection strategies, optimizing surgical techniques, and improving patient surgical safety and postoperative quality of life. In addition, the results of this study also have guiding significance for the innovation and improvement of surgical instruments, which may promote the development of related technologies and equipment, and thus promote their application in a wider range of surgical fields.

ELIGIBILITY:
Inclusion Criteria:

* All cases were the first to undergo open thyroidectomy surgery.
* All clinical data and research materials of the cases are complete.
* All cases underwent thyroid function examination before and after surgery.
* All cases in the experimental group were treated with a head mounted magnifying glass during surgery.

Exclusion Criteria:

* Except for cases of recurrence.
* Cases with incomplete clinical data and research materials are excluded.
* Cases that have not undergone thyroid function tests before and after surgery are excluded.
* Excluding cases of secondary surgery.
* Excluding cases in the experimental group who did not use a head mounted magnifying glass during surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
PTH level | 4 weeks
  To verify the practical effectiveness of wearing a magnifying glass in thyroid surgery, investigators examine changes in PTH levels before and after surgery.
lymph nodes number | 2 weeks
  To verify the practical effectiveness of wearing a magnifying glass in thyroid surgery, investigators follow up on the number of lymph nodes removed in the postoperative pathology report.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided